CLINICAL TRIAL: NCT03614767
Title: Assessment of Predictive Role of Urodynamics in Sacral Neuromodulation Patients
Brief Title: Sacral Neuromodulation & Urodynamics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Donald Vaganée, Principal Investigator, Universiteit Antwerpen
Other Study IDs: 17/30334
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Overactive Bladder; Non-obstructive Urinary Retention
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Urodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successes: Patients with >50% improvement during test procedure of sacral neuromodulation.
  Interventions: Diagnostic Test: urodynamics
- Failures: Patients with <50% improvement during test procedure of sacral neuromodulation.
  Interventions: Diagnostic Test: urodynamics

INTERVENTIONS:
Diagnostic Test: urodynamics — Bladder filling and pressure is measured by the insertion of probes within the bladder, urethra and anorectum.
  Other Names: Ice water test; Slider

SUMMARY:
In the field of urology, sacral neuromodulation (SNM) is a well-accepted, second-line, minimally invasive treatment for patients with overactive bladder dry (OABD) or wet (OABW), and for patients with non-obstructive urinary retention (NOUR).

Long-term vary between 50-60%. This study examines whether urodynamics can be used as a predictor for successful SNM therapy

ELIGIBILITY:
Inclusion Criteria:

* Overactive bladder
* Non-obstructive urinary retention

Exclusion Criteria:

* Neurogenica disorder (e.g. cerebrovascular accident, spinal cord injury)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with overactive bladder or non-obstructive urinary retention.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in bladder volume | 3 weeks
  Change in bladder volume is measured before and after test procedure for sacral neuromodulation
Change in bladder sensation | 3 weeks
  Bladder sensation is measured by a slider (indicating bladder fullness scaled from 0 to 100) before and after test procedure for sacral neuromodulation
Change in ice water test | 3 weeks
  Ice water is infused in the bladder and incontinence upon insertion of the ice water is assessed before and after sacral neuromodulation

CONTACTS AND LOCATIONS:
Overall Officials: Stefan De Wachter, MD PhD FEBU, Study Director — University Hospital, Antwerp
Locations (1):
- University of antwerp, Antwerp, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Undecided